CLINICAL TRIAL: NCT07162155
Title: A Hybrid Program to Prevent Substance Use Risk Among Upper Elementary School Students Using a Positive Youth Development Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Williams (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Christopher Williams, Senior Research Scientist, National Health Promotion Associates, Inc.
Organization: National Health Promotion Associates, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61665-01-2024; R44DA061665 (NIH)
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Vaping; E Cig Use; Prescription Drug Misuse
Keywords: prevention; school-based; positive youth development
MeSH Terms: conditions — Vaping; Prescription Drug Misuse

STUDY DESIGN:
Intervention Model Description: Psychosocial school-based hybrid intervention which includes traditional classroom sessions and online e-learning modules to reduce risk of vaping and prescription drug misuse as part of a broader positive youth development substance use prevention model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classroom Sessions and E-learning Modules (Experimental): Students will: attend 1 classroom session per week for 6 weeks (lecture, discussion, small group activities, skills practice) and complete 1 e-learning module per week for 6 weeks (animated didactic content).
  Interventions: Behavioral: School-based Hybrid Intervention to Prevent Vaping and Prescription Drug Misuse
- Control Condition (No Intervention): Students attending schools randomized to the control group will attend existing health education programming.

INTERVENTIONS:
Behavioral: School-based Hybrid Intervention to Prevent Vaping and Prescription Drug Misuse — Psychosocial school-based hybrid intervention which includes traditional classroom sessions and online e-learning modules to reduce risk of vaping and prescription drug misuse among upper elementary school students.
  Arms: Classroom Sessions and E-learning Modules

SUMMARY:
The goal of this randomized controlled trial is to evaluate a psychosocial school-based hybrid intervention which includes traditional classroom sessions and online e-learning modules to reduce risk of vaping and prescription drug misuse as part of a broader positive youth development substance use prevention model. Upper elementary schools (N=30) will be randomized to either an intervention group that will receive a hybrid intervention or a treatment-as-usual control group that will receive existing health education programming. At the end of the intervention period, and at 6- and 12-month follow-up assessments, both groups will be compared on changes in behaviors, norms, attitudes, and knowledge regarding vaping and prescription medication use.

The main questions the trial aims to answer are:

* Does the intervention lower risk of vaping and prescription drug misuse?
* Does the intervention increase pro-health norms, attitudes, and knowledge regarding vaping and prescription drug misuse?

Participants will:

* Attend 1 classroom session per week for 6 weeks (lecture, discussion, small group activities, skills practice).
* Complete 1 e-learning module per week for 6 weeks (animated didactic content).
* Students attending schools randomized to the control group will attend existing health education programming.

DETAILED DESCRIPTION:
This SBIR Fast-Track proposal is designed to address the urgent problems of vaping and prescription drug misuse (PDM) among youth in the U.S. There is a dearth of primary prevention programs for vaping and PDM that have demonstrated changes in behavior as part of a rigorously designed evaluation. Research shows that the age of onset for these behaviors is decreasing and rates are increasing among the youngest cohorts. While there are a number of substance use prevention programs, there are no evidence-based programs that focus on these problems among upper elementary school students from a positive youth development perspective. Furthermore, due to growing constraints on classroom time, new evidence-based hybrid prevention programs are needed that flexibly incorporate the use of online digital technology and classroom components. In the proposed project, we will develop and test a hybrid adaptation of the evidence-based Life Skills Training (LST) substance abuse prevention program for upper elementary school students. The LST program has been extensively tested and found to effectively prevent substance abuse in a series of randomized controlled trials with behavioral effects reported in over 30 peer-reviewed publications. The proposed hybrid preventive intervention will: 1) utilize both online e-learning modules and traditional classroom sessions to reduce risk of vaping and PDM as part of a broader positive youth development substance use prevention model; 2) teach students about the harms of vaping and the importance of safe and appropriate prescription medication use; 3) enhance protective factors by building social and self-regulation skills through interactive learning and behavioral rehearsal scenarios; and 4) incorporate online booster sessions. In Phase I, we will develop prototypes of e-learning modules and classroom materials and focus group test them with upper elementary school students, teachers, and parents to demonstrate feasibility, relevance, usability, and appeal. Materials will be revised based on focus group feedback and fully developed, and then we will conduct a rigorous national randomized trial of the prevention program in Phase II. Elementary schools (N=30) will be randomized into either an intervention group that will receive the new hybrid intervention or a treatment-as-usual control group that will receive existing health education programming. At the end of the intervention period, and at 6- and 12-month follow-up assessments, we will compare both groups on changes in behaviors, norms, attitudes, and knowledge regarding vaping and appropriate prescription medication use. This research offers the potential to identify an innovative, effective, interactive, and engaging hybrid preventive intervention program that reduces the time burden for classroom prevention by incorporating e-learning modules as part of an evidence-based prevention model. The intervention materials may help to reduce risk for emergent substance use behaviors among upper elementary school youth. The program can be widely disseminated throughout the country and ultimately decrease the harms of substance misuse among youth.

ELIGIBILITY:
Inclusion Criteria: Students will be eligible for participation if they attend a school enrolled in the trial and they are between ages 7-11.

Exclusion Criteria: All students will be eligible to participate in intervention implmentation, but survey responses will be excluded from the formal analysis with documentation of significant cognitive impairment as determined by school officials.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Vaping, e-cigarette use, and prescription drug misuse behaviors, norms, and attitudes at baseline | Pre-test (prior to participating in the first session/module of the intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding vaping, e-cigarette use, and prescription drug misuse behaviors and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline baseline vaping, e-cigarette, and prescription drug misue behaviors, norms, and attitudes at post-intervention | Post-test (within 2 weeks of completing final session/module of the intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding vaping, e-cigarette use, and prescription drug misuse behaviors and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in bse line vaping, e-cigarette use, and prescription drug misuse behaviors, norms, and attitudes at 6-month followup | 6-month followup (within-in 6-7 months of completing final session of interventioon)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding vaping, e-cigarette use, and prescription drug misuse behaviors and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline vaping, e-cigarette use, and prescription drug misuse behaviors, norms, and attitudes at 12-month followup | 12-month followup (within 12-13 months of completing final session of intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding vaping, e-cigarette use, and prescription drug misuse behaviors and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- National Health Promotion Associates, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No